CLINICAL TRIAL: NCT06594172
Title: A Phase II Clinical Trial of of Early Application of Memantine and Pioglitazone to Protect Cognitive Function After Radiotherapy
Brief Title: Early Application of Memantine and Pioglitazone to Protect Cognitive Function After Radiotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Fujian Medical University Union Hospital (Other); Southern Medical University, China (Other); The Affiliated Panyu Center Hospital of Guangzhou Medical University (Unknown); The Central Hospital of Shaoyang City (Unknown)
Responsible Party: Principal Investigator, Yuan yawei, The Chair of the Department of Radiation Oncology, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMUCR2024-01019
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Radiation Disease; Cognitive Impairment; Drug Effect
Keywords: radiation induced brain injury; Memantine; Pioglitazone; cognitive function
MeSH Terms: conditions — Abnormalities, Radiation-Induced; Cognitive Dysfunction | interventions — Memantine; Pioglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MPR (Experimental): combined Memantine and Pioglitazone with radiation therapy
  Interventions: Drug: Memantine Oral Tablet; Drug: Pioglitazone 15mg; Radiation: Hippocampal avoidance whole-brain radiotherapy (HA-WBRT)

INTERVENTIONS:
Drug: Memantine Oral Tablet — Oral administration of Memantine Tablets (10mg/tablet):
  Week 1: 5mg in the morning. Week 2: 5mg twice daily. Week 3: 10mg in the morning, 5mg in the evening. Weeks 4-24: 10mg twice daily.
  Other Names: pioglitazone; hippocampal avoidance whole-brain radiotherapy (HA-WBRT)
Drug: Pioglitazone 15mg — Simultaneous oral administration of Pioglitazone Tablets (15mg/tablet):
  Weeks 1-24: 30mg once daily.
Radiation: Hippocampal avoidance whole-brain radiotherapy (HA-WBRT) — Based on the RTOG 0933 protocol, hippocampal and perihippocampal regions are delineated, and hippocampal dose constraints are applied. The radiation dose to the perihippocampal region is determined based on the size, number, and volume of brain metastases (whole-brain radiation therapy: DT 30Gy/10F, weeks 1-2; with a simultaneous boost to the pathological local area if necessary, 10-20Gy).

SUMMARY:
This clinical trial aims to evaluate the efficacy of early intervention with Memantine and Pioglitazone in preventing Radiation-Induced Brain Injury (RIBI) in patients undergoing cranial radiotherapy.

RIBI, a significant complication of radiation therapy for primary and metastatic brain tumors, as well as head and neck cancers, often presents with delayed and irreversible neurological damage, severely affecting patients' quality of life.

Our previous studies have indicated that Memantine, an NMDAR antagonist, and Pioglitazone, a PPAR-γ agonist, play crucial roles in modulating the neuroprotective immune microenvironment by targeting key mechanisms of neuron-astrocyte fatty acid metabolism coupling. These findings suggest that early administration of these drugs could protect cognitive function and reduce neuroinflammation in patients post-radiation.

This prospective phase II clinical trial will assess the combined efficacy of Memantine and Pioglitazone in improving cognitive outcomes and preventing RIBI without adversely impacting the anti-tumor efficacy of radiation therapy. The study will also explore the synergistic effects of these two FDA-approved drugs in early-stage RIBI prevention, providing a new therapeutic strategy for enhancing the quality of life in cancer patients receiving radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Recursive Partitioning Analysis (RPA), Class I ~ Class II
* Karnofsky Performance Status of ≥70
* The primary tumor must be pathologically confirmed. For newly diagnosed brain metastases, the number of metastases is not limited, but the brain metastases could not have been within 5 mm of hippocampus. Additionally, there must be no hard or soft meningeal metastases.
* No history of whole-brain radiation therapy; patients who are eligible for surgical resection of brain metastases prior to radiation therapy are allowed.
* Bone marrow function: White blood cell count ≥ 4 × 10⁹/L, hemoglobin ≥ 90 g/L, and platelet count ≥ 100 × 10⁹/L.
* Adequate hepatic function: Total bilirubin ≤ 1.5 × ULN (Upper Limit of Normal); ALT (alanine aminotransferase), AST (aspartate aminotransferase) ≤ 2.5 × ULN; ALP (alkaline phosphatase) ≤ 2.5 × ULN and total bilirubin ≤ ULN.
* Adequate renal function: creatinine clearance rate ≥ 30 ml/min.
* Patients or their legal guardians voluntarily participate and sign the informed consent form.

Exclusion Criteria:

* Radiographic evidence of hydrocephalus or other architectural distortion of the ventricular system, including placement of external ventricular drain or ventriculoperitoneal shunt.
* Planned cytotoxic chemotherapy during the WBRT.
* Pregnant or lactating women (Women of childbearing age must undergo a pregnancy test; effective contraception must be enforced during the treatment period).
* Previous cranial radiation therapy (Except for patients with head and neck cancer where the disease site is outside the cranial radiation field).
* Severe or active symptomatic cardiopulmonary diseases; clinically significant psychiatric disorders; Personality or psychiatric disease; Severe hepatic disease defined as a diagnosis of Child-Pugh class B or C hepatic disease;
* Intolerant to or allergic to Memantine or pioglitazone.
* Difficulty swallowing, chronic diarrhea, or bowel obstruction.
* NYHA class III or IV heart failure or symptomatic peripheral edema (grade 2 or higher); those treated with insulin or oral hypoglycemic agents for steroid-induced hyperglycemia, or those currently using other NMDA antagonists.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
the cumulative incidence of cognitive failure | At weeks 4, 8, 16, 24, 36, and 48 after the completion of radiotherapy
  the proportion of participants who experience cognitive impairments after radiation therapy

SECONDARY OUTCOMES:
Cognitive Score Decline | At weeks 4, 8, 16, 24, 36, and 48 after the completion of radiotherapy
  based on the Reliable Change Index of at least one cognitive test
Progressive-free survival for Intracranial Tumors | At weeks 4, 8, 16, 24, 36, and 48 after the completion of radiotherapy
  latencies to the first intracranial treatment failure or death from any cause
Overall Survival | At weeks 4, 8, 16, 24, 36, and 48 after the completion of radiotherapy
  death due to any cause